CLINICAL TRIAL: NCT00176007
Title: Hypoxia Impairs Systemic Endothelial Function in Individuals Prone to High-Altitude Pulmonary Edema.
Brief Title: Hypoxia Impairs Endothelial Function in HAPEs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: A001
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Healthy

INTERVENTIONS:
Procedure: Hypoxia

SUMMARY:
Aim of the study is to investigate the function of the systemic vascular endothelium in individuals susceptible to high-altitude pulmonary oedema during normoxia and normobaric hypoxia.

DETAILED DESCRIPTION:
Rationale: High-altitude pulmonary edema (HAPE) is characterized by excessive pulmonary vasoconstriction and is associated with decreased concentrations of nitric oxide (NO) in the lung. Objectives: We hypothesized that individuals susceptible to HAPE (HAPE-S) would also have dysfunction of the vascular NO vasodilator pathway during hypoxia in the systemic vasculature. Methods: During normoxia (FI(O(2)) = 0.21) and 4 hours of normobaric hypoxia (FI(O(2)) = 0.12, corresponding to an altitude of 4,500 m above sea level) endothelium-dependent and endothelium-independent vasodilator responses to intraarterial infusion of acetylcholine (ACh) and sodium nitroprusside, respectively, were measured by forearm venous occlusion plethysmography in nine HAPE-S subjects and in nine HAPE-resistant control subjects. Main Results: Pulmonary artery systolic pressure increased from 22 +/- 3 to 33 +/- 6 mm Hg (p < 0.001) during hypoxia in control subjects, and from 25 +/- 4 to 50 +/- 9 mm Hg in HAPE-S subjects (p < 0.001). Despite similar responses during normoxia in both groups, ACh-induced changes in forearm blood flow markedly decreased during hypoxia in HAPE-S subjects (p = 0.01) but not in control subjects. The attenuated vascular response to ACh infusion during hypoxia inversely correlated with increased pulmonary artery systolic pressure (p = 0.04) and decreased plasma nitrite correlated with attenuated ACh-induced vasodilation in HAPE-S subjects (p = 0.02). Conclusions: Hypoxia markedly impairs vascular endothelial function in the systemic circulation in HAPE-S subjects due to a decreased bioavailability of NO. Impairment of the NO pathway could contribute to the enhanced hypoxic pulmonary vasoconstriction that is central to the pathogenesis of HAPE.

ELIGIBILITY:
Inclusion Criteria:

Healthy, male volunteers, age: 18-55

- Able and willing to give written informed consent

Exclusion Criteria:

* Known condition causing endothelial dysfunction (e.g. diabetes, hyperlipidaemia, arterial hypertension, smoking, hyperhomocysteinaemia)
* Regular medication and/or treatment with drugs within the last 4 weeks (exclusion has to be decided in each case)
* Acute or chronic illness
* Participation in clinical trial/blood donation within 2 month before the study
* Nicotine, drug and/or alcohol abuse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Haefeli, MD, Principal Investigator — Heidelberg University